CLINICAL TRIAL: NCT00260481
Title: Double-Blind, Placebo Controlled Trial of Prometa Pharmacotherapy for the Treatment of Methamphetamine Abuse
Brief Title: Prometa Pharmacotherapy for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Walter Ling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-01-076-01
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Drug Abuse; Drug Dependence
Keywords: Methamphetamine Dependence; Pharmacotherapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): During the Infusion periods, participants in the placebo condition will receive pre-treatment with hydroxyzine (50mg) followed by placebo medications administered both orally and through infusion, as well as a second dose of hydroxyzine (50mg), delivered at the same rate and delivery system to match the active condition. All participants may receive daily multivitamins as determined appropriate by the study physician. Multivitamins are not considered active medications for the PROMETA pharmacotherapy, but may be provided to participants in both conditions at the same rates and delivery methods for the duration of the study. Because participants are treatment-seeking and use of a placebo condition is warranted, all participants will be provided with once weekly, manual-guided cognitive behavioral therapy sessions during all outpatient periods of the study.
  Interventions: Drug: Placebo
- Prometa (Active Comparator): During the infusion periods, participants assigned to the PROMETA pharmacotherapy condition will receive pre-treatment with hydroxyzine (50mg) followed by intravenous flumazenil (2mg) over a 2-hour period. Before bedtime, patients will again take 50mg of hydroxyzine orally, as well as 300mg of oral gabapentin (participants will titrate up their dosage of gabapentin each day - 300mg on day 0, 600mg on day 1, 900mg on day 2). All participants may receive daily multivitamins as determined appropriate by the study physician. Multivitamins are not considered active medications for the PROMETA pharmacotherapy, but may be provided to participants in both conditions at the same rates and delivery methods for the duration of the study. Because participants are treatment-seeking and use of a placebo condition is warranted, all participants will be provided with once weekly, manual-guided cognitive behavioral therapy sessions during all outpatient periods of the study.
  Interventions: Drug: Prometa

INTERVENTIONS:
Drug: Prometa — Medication protocol includes 2 infusion periods of 3 and 2 days, respectively and outpatient medications for 39 days
  Arms: Prometa
Drug: Placebo — Placebo protocol includes 2 infusion periods of 3 and 2 days, respectively and outpatient placebo medications for 39 days.
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess the efficacy of the PROMETA pharmacotherapy compared to placebo for initiating abstinence and for preventing relapse to methamphetamine use in treatment-seeking individuals meeting criteria for methamphetamine abuse. It is hypothesized that individuals assigned to receive the PROMETA pharmacotherapy, compared to placebo, will demonstrate significantly fewer and less intense withdrawal symptoms, more days abstinent from methamphetamine use, and fewer relapses to methamphetamine use as assessed by self-report of drug use verified by urine samples.

DETAILED DESCRIPTION:
Using a double-blind placebo design, the effectiveness of the Prometa protocol for methamphetamine dependence will be investigated as compared to a placebo condition. The procedure utilizes a combination of medications delivered both orally and by infusion in a controlled medical setting. Participants will be randomly assigned to the active medication or placebo condition, and will receive medications for 40 days, including two inpatient hospitalization phases of three days each. All participants will also receive once-weekly psychosocial cognitive-behavioral therapy throughout the 106 day study duration. A variety of data will be collected throughout the study, including psychological, cognitive, medical, and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years-of-age;
* Have a DSM-IV-TR diagnosis of methamphetamine abuse or dependence as determined by SCID;
* Be seeking treatment for methamphetamine abuse or dependence;
* Be able to understand, and having understood, provide written informed consent;
* If female and of child bearing potential, agree to use an approved method of birth control or be surgically sterile;
* Have completed all other psychological assessments; -Have used methamphetamine at least 4 of the last 30 days. -

Exclusion Criteria:

* Have current dependence, defined by DSM-IV-TR criteria, on any psychoactive substance other than methamphetamine, alcohol, nicotine, or marijuana or physiological dependence on alcohol requiring medical detoxification (CIWA-AR score ≥ 15);
* Be mandated by the court to obtain treatment for methamphetamine-abuse or dependence;
* Be anyone who, in the opinion of the investigator, would not be expected to complete the study protocol due to probable incarceration or relocation from the clinic area;
* Have a current or previous psychiatric, or a neurological disorder including but not limited to epilepsy and absence seizures, fainting spells, brain disease, dementia, or any disorder that, in the opinion of the study physician requires ongoing treatment that would make study participation unsafe or which would make treatment compliance difficult.
* Have a psychiatric disorder, as assessed by the SCID, or a neurological disorder including but not limited to epilepsy and absence seizures, brain disease, dementia or any disorder that, in the opinion of the study physician, requires ongoing treatment that would make study participation unsafe or which would make treatment compliance difficult;
* Have had electroconvulsive therapy within the past 3 months preceding screening; Have current suicidal ideation or plan (within the past 30 days) as assessed by the SCID;
* Be pregnant or lactating;
* Have serious medical illnesses (including, but not limited to: uncontrolled hypertension, significant heart disease including myocardial infarction within one year of enrollment, or any clinically significant cardiovascular abnormality (ECG), hepatic, renal or gastrointestinal disorders that could result in a clinically significant alteration of metabolism or excretion of the study agent, potentially life-threatening or progressive medical illness other than addiction that may compromise subject safety or study conduct);
* Have clinically significant abnormal laboratory values;
* Benzodiazepine and/or similar sedative-hypnotic or anxiolytic use or abuse within 15 days of potential PROMETA Treatment;
* Must not be habituated to benzodiazepines and must provide a urine sample that is negative for benzodiazepines;
* Must not be taking supra-therapeutic doses of zolpidem (Ambien TM) or zaleplon (Sonata TM); Taking clonazepam (Klonopin TM) or other benzodiazepine;
* Patients must not be taking cyclic antidepressants, lithium, methylxanthines, isoniazid, propoxyphene, monoamine oxidase inhibitors, buproprion HCL, and cyclosporine.
* Have AIDS;
* Have active tuberculosis (positive tuberculin test and confirmatory diagnostic chest x-ray);
* Have known or suspected hypersensitivity to PROMETA;
* Have been treated with PROMETA for any reason currently or during the past year;
* Have any disorder or condition that, in the opinion of the study physician, would make study participation difficult or unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Abstinence across the duration of the study | from screening to termination

SECONDARY OUTCOMES:
Days of methamphetamine use | from screening to termination
days of other drug use | from screening to termination
cognitive functioning | comparison of pre- to post-treatment scores

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — UCLA Integrated Substance ABuse Programs
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States

REFERENCES:
- [Derived] Ling W, Shoptaw S, Hillhouse M, Bholat MA, Charuvastra C, Heinzerling K, Chim D, Annon J, Dowling PT, Doraimani G. Double-blind placebo-controlled evaluation of the PROMETA protocol for methamphetamine dependence. Addiction. 2012 Feb;107(2):361-9. doi: 10.1111/j.1360-0443.2011.03619.x. Epub 2011 Nov 15. PMID 22082089